CLINICAL TRIAL: NCT05198206
Title: Current Status of Diagnosis and Treatment of Pregnancy With Pulmonary Hypertension and Maternal and Infant Outcomes: a Multicentre Retrospective Study in China
Brief Title: Pregnant Women With Pulmonary Hypertension in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wei Huang, Professor Wei Huang, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2021XMSB0011013
Record Dates: First submitted 2021-11-13; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Hypertension; Pregnancy, High Risk
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (32):
- The First Affiliated Hospital of Chongqing Medical University
- West China Hospital
- the First Affiliated Hospital of Xi'an Jiaotong University
- Guangdong Provincial People's Hospital
- Xiangya Hospital of Central South University
- The Second Affiliated Hospital of Harbin Medical University
- Yan'an Hospital of Kunming City
- Zhongshan Hospital
- Gansu Provincial People's Hospital
- Qilu Hospital of Shandong University
- Shanxi Provincial Cardiovascular Hospital
- West China Second Hospital
- The First Affiliated Hospital of Jilin University
- Xinqiao Hospital, Army Medical University
- The First Affiliated Hospital of Guangzhou Medical University
- the Second Xiangya Hospital of Central South University
- Shengjing Hospital of China Medical University
- The Second Affiliated Hospital of Nanchang University
- Henan Provincial People's Hospital
- Southwest Medical University Hospital
- The First Affiliated Hospital of Gannan Medical University
- University-town Hospital of Chongqing Medical University
- Chongqing Health Center for Women and Children
- Kunhua Hospital
- Changdu People's Hospital of Tibet
- The Sixth People's Hospital of Chengdu
- Chongqing Bishan District People's Hospital
- Sichuan Guangyuan People's Hospital
- Xinjiang Military Region General Hospital
- Xinjiang Uygur Autonomous Region People's Hospital
- The First Affiliated Hospital of Anhui Medical University
- Yantai Yuhuangding Hospital

SUMMARY:
Little is known about the status of maternal, obstetric and neonatal complications and the potential predictors of developing heart failure (HF) in the mothers with pulmonary hypertension in China. Eligible samples were screened from January, 2012 to December, 2021. Maternal clinical characteristics and in-and-out hospital outcomes were collected and compared in women with and without pulmonary hypertension.

The main aims of this study are as follows:

1. To investigate the perinatal diagnosis and treatment of pregnant women with pulmonary hypertension in China over the past 10 years and the maternal and infant outcomes.
2. To explore risk factors that affect the outcome of pregnant women with pulmonary hypertension in mothers and infants.
3. To summarise effective risk stratification management protocols and construct standardised strategies for the management of pulmonary hypertension in pregnancy.
4. To establish a clinical database, biobank and follow-up cohort for pregnant women with pulmonary hypertension across China.

DETAILED DESCRIPTION:
Pulmonary hypertension is a malignant disease with a high mortality rate, difficult to diagnose at an early stage and has posed a huge economic burden on patients and society. Pregnancy with pulmonary hypertension is associated with high maternal mortality (25% - 56% ) and a high incidence of fetal complications such as preterm birth (85% - 100%), fetal growth restriction (3% - 33%) and severe outcomes such as fetal/neonatal loss (7% - 13%). A high maternal mortality rate of 30%-56% for pregnancy-related pulmonary hypertension for women and 11-28% for infants has been reported.

However, despite national and international guidelines recommending avoidance of pregnancy, some women with pulmonary hypertension persist in their pregnancies or have unplanned pregnancies, and some pregnant women are diagnosed with pulmonary hypertension only after symptoms such as heart failure have worsened. Although with the development of pulmonary arterial hypertension(PAH)-targeted drugs, the mortality rate for pregnancy-associated PAH has declined but remains relatively high. The high maternal and infant mortality rates and complication rates make it a critical condition that seriously endangers the lives of both mother and child.

Limited data in China reported the outcome, prognosis and management measures of combined pulmonary hypertension in pregnancy, and there is a lack of overall description and analysis of pregnancy with pulmonary hypertension in a multi-centre setting. The current status of high risk factors, efficacy of multidisciplinary consultation and management of maternal and fetal mortality and complications is unclear.

Therefore, the aim of this study was to retrospectively analyse the current status of the management of pregnant women with pulmonary hypertension in a multicenter setting across China, and try to summarise effective risk stratification management protocols and construct standardised strategies for the management of pulmonary hypertension in pregnancy to reduce maternal and infant mortality and adverse events and improve the prognosis of mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women, regardless of age, race
* diagnosed with pulmonary hypertension(PH) before pregnancy or during pregnancy
* diagnosed with PH by right heart catheterization or echocardiography
* diagnostic criteria of right heart catheterization: mean pulmonary artery pressure (mPAP) ≥ 25 mm Hg by right heart catheterization at rest
* diagnostic criteria of echocardiography: pulmonary artery systolic pressure (PASP)≥40 mm Hg
* time: from January 1, 2012 to December 31, 2021

Exclusion Criteria:

* Patients with isolated exercise-induced PH (mean PAP <25 mm Hg at rest and >30 mm Hg at exercise) were excluded.
* pulmonary artery systolic pressure (PASP)<40 mmHg by echocardiography
* mean pulmonary artery pressure (mPAP) < 25 mm Hg by right heart catheterization at rest

Ages: 14 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregant women who conform to echocardiographic or right heart catheter criteria of PAH in 32 centers across China were included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
all-cause maternal mortality | diagnosis of pregnancy to six months postpartum in 2012-2021
  Investigating the maternal mortality rate from the diagnosis of pregnancy to six months postpartum

SECONDARY OUTCOMES:
Maternal incidence of cardiovascular complications | from diagnosis of pregnancy to six months postpartum in 2012-2021
  heart failure ,arrhythmias, thrombotic events (including valve thrombosis) , aortic dissection and other cardiovascular complications during pregnancy until 6 months postpartum
the incidence of obstetric events | From delivery to 42 days postpartum
  the incidence of post-partum hemorrhage, emergency Caesarean section, pre-eclampsia, eclampsia or pregnancy-induced hypertension From delivery to 42 days postpartum
the incidence of fetal events | From delivery to 42 days postpartum
  prematurity , fetal mortality, early neonatal mortality, intra-uterine growth retardation, low birth weight or low Apgar score from delivery to 42 days postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes